CLINICAL TRIAL: NCT04668053
Title: Effects of Hip Flexor Resistance Training On Strength, Speed and Agility in Young Female Cricket Players
Brief Title: Hip Flexor Resistance Training on Pin Young Female Cricket Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00578 Saima Naseem
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Hip Flexion Contractures
Keywords: Agility; Hip flexors; Resistance training; Speed; strength
MeSH Terms: conditions — Hip Contracture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional training protocol (Active Comparator): Mobility and core strengthening, The step, The Lunge, Body weight squat, Body weight split squat , Bilateral hip raise, Push-up ,Cricket related skills
  Interventions: Other: Traditional training protocol
- Hip flexor resistance protocol (Experimental): Mobility and core strengthening, The step, The Lunge, Body weight squat, Body weight split squat , Bilateral hip raise, Push-up ,Cricket related skills and hip flexors resistance protocol
  Interventions: Other: Hip flexor resistance protocol

INTERVENTIONS:
Other: Traditional training protocol — Mobility and core strengthening and the steps and lunges As per athletes requirement Body weight squat with 12 reps, Body weight split squat with 8 each side, Bilateral hip raise with 12 reps, Push-up with15 reps and Cricket related skills as per coach advised
  Arms: Traditional training protocol
Other: Hip flexor resistance protocol — Warm up prior to training The loop bands (Resistance-band©) that were used are in several colors-Red, black, yellow, blue and green extended from strongest type to weakest.
  Athletes executed 3 training sessions of 3 sets per week for 6 weeks.
  The relative load was:
  Week 1----15 RM Week 2-4----10 RM Week 5-6----8 RM The Therapist has ensured a concentric contraction of 3-s, an isometric contraction of 2-s, eccentric contraction of 3-s, rest for 2-s prior to the next repetition and rest for 2-min prior the next set.
  It took 10 min to complete each session, with rest between sets.
  Arms: Hip flexor resistance protocol

SUMMARY:
The aim of this research is to study the role of hip flexor strength in the act of particular movement tasks generally required in cricket. In young cricket players, hip flexor training protocol may be productive in improving the acceleration time of sprint and shuttle run.

It was a Randomized Controlled Trial conducted in National Cricket Academy Lahore, Lahore zonal Cricket Academy, Multan High Performance Cricket Centre during 6 months. 30 participants were selected through Non Probability Convenience Sampling Technique with inclusion criteria Female cricket players involved in their training programs aged 17-25 years and Participants should be bodily active before the start of trial for minimum 30 minutes a day for 5 days of week. The participants were excluded if Systematic strength training Performed by the athletes for the hip flexors more than a week before the start of trial and if Athlete suffered an injury or having pain in low back area, hips or lower limbs in last 6 months or if they have any diagnosed Neuro-musculoskeletal, musculo-skeletal pathology. The Data Collection Tools were 40-yd Dash Test, Shuttle Run and Dynamometer.

DETAILED DESCRIPTION:
Cricket has undergone dramatic changes in recent years, with the development of one day and Twenty-twenty cricket altering some of the vital characteristics of the game. The shorter game formats tend to be more physically intensive when related to match duration, incorporating more maximal sprints when fielding, bowling, and batting. As a result of these demands, running speed has become an essential athletic quality for cricketers and therefore must be assessed correctly. Based on the action of the legs, a running cycle can be subdivided into 3 phases-a supporting phase that begins when the foot lands and ends when the athlete's center of gravity (CG) passes forward of it, a driving phase that begins as the supporting phase ends and ends as the foot leaves the ground, and a recovery phase during which the foot is off the ground and is being brought forward preparatory to the next landing. Although quadriceps, hamstrings, and calf muscles are mainly responsible for propelling the body forward during running and jumping exercises, hip flexor muscles also contribute to these actions. Specifically, the hip flexor muscles assist in bringing the free leg forward and upward during the recovery phase of running. Muscular strength is one of the components of physical fitness. Athletes of different sports use resistance training to improve their muscular strength. Among the exercises that are commonly performed by athletes, hip flexion is one of the most ignored exercises in strength and conditioning for sports performance. Hip flexion exercises are often neglected in strength training programs for popular sports such as football, basketball, and soccer. Young et al. in 2011 study of the effects of strength training and reported that 2 sessions per week over a soccer season produced significant gains in isokinetic hip flexor and extensor strength as well as knee extensor and flexor strength. This was accompanied by a significant increase in maximum kicking distance, which was not observed in non-strength trained players. F. Tyler et al reported that the hip strength and flexibility play role in the incidence of adductor and hip flexor strains in ice hockey players. Deane et al. in an RCT compares two types of training programs, it was observed that high resistance training resulted in an improved initial acceleration phase, whereas high-velocity training resulted in an improved initial acceleration and maximum speed. Almost all methods or interventions focus on muscles associated with the driving phase of running (i.e., gluteus maximus, 2 quadriceps, and plantar flexors), whereas the training of muscles responsible for the recovery phase has not been explored. Specific ways of strengthening the hip-flexors in injury prevention or post-surgical rehabilitation have not previously been well described in the sports medicine literature. Acute injuries to the rectus femoris are often experienced in kicking sports, such as in the different football codes, whereas longstanding iliopsoas-related pain is common in football players, runners and dancers. Simple ways of improving hip flexor strength and function are needed in injury prevention. In addition to exercise machines and free-weight exercises, resistance training using elastic tubing has been demonstrated to be effective in strength development and improving sports performance. The clinical advantage of the elastic band is that it is portable and inexpensive, takes up very little space and can be used everywhere, indoor as well as outdoor, wherever solid attachment of the elastic band is possible. Hip flexor injuries are common in cricket players.

Literature is available on hip flexor training on soccer and ice hockey and mostly studies are done on the dominant sided leg. This study will be an initial attempt in Pakistan to explore the role of hip flexor strength in the performance of selected movement tasks commonly required in cricket.

ELIGIBILITY:
Inclusion Criteria:

* Female cricket players involved in their training programs
* BMI 18-25
* Participants should be bodily active before the start of trial for minimum 30 minutes a day for 5 days of week.

Exclusion Criteria:

* Systematic strength training Performed by the athletes for the hip-flexors more than a week before the start of trial
* Athlete suffered an injury or having pain in low back area, hips or lower limbs in last 6 months
* Any diagnosed Neuro-musculoskeletal, musculo-skeletal pathology

Ages: 17 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Female cricket players involved in their training programs as of objective and population target.
Enrollment: 60 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
Hand Held Dynamometer: | 6th week
  Muscle testing was performed using the ''make test'' method of muscle testing in which the subject applied a maximum muscle contraction to the examiner's hand holding the dynamometer. Players were asked to hold the muscle contraction for 2 s. The maximum highest force from two trials has been used for strength assessments.

SECONDARY OUTCOMES:
40-yard Dash | 6th week
  This test used to evaluate the acceleration and speed characteristics of an athlete. Participants has been asked to perform a 40-yard sprint from a motionless place which has been used to estimate the acceleration and speed attributes of participant. Each participant executed 2 best effort sprints of 40-yard wearing their own running shoes.
  Time was measured using a digital stop watch
Shuttle Run | 6th week
  20m Shuttle run was used to measure the agility of an athlete. The participants have been requested to Run from side to side between the marked lines of 20 m twice with the maximum effort. Each participant performed 2 runs, and digital stop watch was used to record the completion time

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, MSPT-OMPT, Principal Investigator — Riphah International University
Locations (1):
- National Cricket Academy Lahore, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deane RS, Chow JW, Tillman MD, Fournier KA. Effects of hip flexor training on sprint, shuttle run, and vertical jump performance. J Strength Cond Res. 2005 Aug;19(3):615-21. doi: 10.1519/14974.1. PMID 16095411
- [Background] Petersen CJ, Pyne D, Dawson B, Portus M, Kellett A. Movement patterns in cricket vary by both position and game format. J Sports Sci. 2010 Jan;28(1):45-52. doi: 10.1080/02640410903348665. PMID 20013461
- [Background] Lockie RG, Callaghan SJ, Jeffriess MD. Analysis of specific speed testing for cricketers. J Strength Cond Res. 2013 Nov;27(11):2981-8. doi: 10.1519/JSC.0b013e31828a2c56. PMID 23439342
- [Background] Foran B. High-performance sports conditioning: Human kinetics; 2001.
- [Background] Young WB, Rath DA. Enhancing foot velocity in football kicking: the role of strength training. J Strength Cond Res. 2011 Feb;25(2):561-6. doi: 10.1519/JSC.0b013e3181bf42eb. PMID 20375741
- [Background] Tyler TF, Nicholas SJ, Campbell RJ, McHugh MP. The association of hip strength and flexibility with the incidence of adductor muscle strains in professional ice hockey players. Am J Sports Med. 2001 Mar-Apr;29(2):124-8. doi: 10.1177/03635465010290020301. PMID 11292035
- [Background] Ekstrand J, Hagglund M, Walden M. Epidemiology of muscle injuries in professional football (soccer). Am J Sports Med. 2011 Jun;39(6):1226-32. doi: 10.1177/0363546510395879. Epub 2011 Feb 18. PMID 21335353
- [Background] Holmich P. Long-standing groin pain in sportspeople falls into three primary patterns, a "clinical entity" approach: a prospective study of 207 patients. Br J Sports Med. 2007 Apr;41(4):247-52; discussion 252. doi: 10.1136/bjsm.2006.033373. Epub 2007 Jan 29. PMID 17261557
- [Background] Werner J, Hagglund M, Walden M, Ekstrand J. UEFA injury study: a prospective study of hip and groin injuries in professional football over seven consecutive seasons. Br J Sports Med. 2009 Dec;43(13):1036-40. doi: 10.1136/bjsm.2009.066944. PMID 19945984
- [Background] Thorborg K, Bandholm T, Zebis M, Andersen LL, Jensen J, Holmich P. Large strengthening effect of a hip-flexor training programme: a randomized controlled trial. Knee Surg Sports Traumatol Arthrosc. 2016 Jul;24(7):2346-52. doi: 10.1007/s00167-015-3583-y. Epub 2015 Mar 22. PMID 25796586